CLINICAL TRIAL: NCT07092462
Title: The Impact of Doomscrolling and Social Media Dependency on Individuals Suffering From Fibromyalgia. A Cross-Sectional Study
Brief Title: Fibromyalgia and the Act of Scrolling Through Social Media.
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Collaborators: Balikesir University (Other)
Responsible Party: Principal Investigator, Faika SANAL KARAHAN, Principal Investigator, Uşak University
Other Study IDs: UsakPDR
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia; Social Media Addiction
Keywords: fibromaylgia; doomscrolling; sleep disturbances; quality of life
MeSH Terms: conditions — Fibromyalgia; Internet Addiction Disorder; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia patients: individuals suffering from fibromyalgia
- Healthy subjects: healthy subjects will be matched with controls demographically (age, gender and education).

SUMMARY:
In recent years, the widespread use of social media and digital platforms has led to the emergence of behavioural patterns such as doomscrolling, which involves the compulsive consumption of negative or distressing online content. This can often lead to increased anxiety and psychological distress. While this phenomenon has been studied extensively in the general population, its impact on individuals with chronic pain conditions, particularly fibromyalgia, remains largely unexplored. FM is a complex disorder characterised by widespread musculoskeletal pain, fatigue, sleep disturbances and cognitive difficulties, often accompanied by heightened emotional distress. As FM patients often experience anxiety and depression and engage in maladaptive coping strategies, doomscrolling may exacerbate their symptoms and impair their overall well-being.

Existing research suggests that excessive social media use is linked to social media addiction (SMA), fear of missing out (FoMO) and poor sleep quality - all of which are particularly relevant to FM patients, who already struggle with sleep dysfunction and psychosocial challenges. Nevertheless, no investigation heretofore has specifically scrutinised the association between doomscrolling, SMA, FoMO and fibromyalgia-related disability. Understanding these associations could provide valuable insights into how digital behaviours influence FM symptomatology and help to identify potential intervention targets to mitigate negative outcomes.

DETAILED DESCRIPTION:
In recent years, the widespread use of social media and digital platforms has led to the emergence of behavioural patterns such as doomscrolling, which involves the compulsive consumption of negative or distressing online content. This can often lead to increased anxiety and psychological distress. While this phenomenon has been studied extensively in the general population, its impact on individuals with chronic pain conditions, particularly fibromyalgia, remains largely unexplored. FM is a complex disorder characterised by widespread musculoskeletal pain, fatigue, sleep disturbances and cognitive difficulties, often accompanied by heightened emotional distress. As FM patients often experience anxiety and depression and engage in maladaptive coping strategies, doomscrolling may exacerbate their symptoms and impair their overall well-being.

Existing research suggests that excessive social media use is linked to social media addiction (SMA), fear of missing out (FoMO) and poor sleep quality - all of which are particularly relevant to FM patients, who already struggle with sleep dysfunction and psychosocial challenges. Nevertheless, no investigation heretofore has specifically scrutinised the association between doomscrolling, SMA, FoMO and fibromyalgia-related disability. Understanding these associations could provide valuable insights into how digital behaviours influence FM symptomatology and help to identify potential intervention targets to mitigate negative outcomes.

This cross-sectional study aims to: - assess the prevalence and severity of doomscrolling in fibromyalgia patients;- examine the relationships between doomscrolling, social media addiction (Bergen Scale), fear of missing out (FoMO Scale), fibromyalgia impact (Fibromyalgia Impact Questionnaire) and sleep disturbances (Pittsburgh Sleep Quality Index);- explore whether doomscrolling and related digital behaviours are associated with worse fibromyalgia symptom severity and quality of life.

By investigating these associations, the study will contribute to the growing body of literature on digital well-being in populations with chronic pain and inform future interventions aimed at promoting healthier media consumption habits among patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Being within the 18-49 age group (based on date of birth).
* Not practising any regular sport or exercise.
* Not having any chronic health problems or physical disabilities.
* Volunteering to participate in the study.

Exclusion Criteria:

* The presence of diagnosed neurological diseases that may adversely affect quality of life (similar to MS or migraine).
* The presence of diagnosed psychiatric diseases that may adversely affect quality of life (similar to depression or OCD).
* The presence of diagnosed rheumatological diseases that may adversely affect quality of life (e.g. rheumatoid arthritis or ankylosing spondylitis).
* Not using a smartphone as part of one's lifestyle (i.e. not using applications).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * The sample will consist of patients diagnosed with "Fibromyalgia" who are under the follow-up of Uşak Training and Research Hospital, Department of Physical Medicine and Rehabilitation.
  * A small control group of 50 participants will be included in the study. To minimise confounding factors, healthy subjects will be matched with controls demographically (age, gender and education).
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Doomscrolling Scale | Baseline
  Sharma et al. developed the Doomscrolling Scale to measure the extent to which participants scroll through persistently negative information on social media.
  Satıcı et al. conducted a study to create a Turkish version of the scale. The scale consists of 15 items. It is a 7-point Likert scale, where 1 equals strongly disagree and 7 equals strongly agree. High scores imply high levels of doomscrolling.
  In this study, the scale will be used with adults.
Bergen Social Media Addiction Scale | Baseline
  The Bergen Social Media Addiction Scale (BSMAS) will be used by the researchers to assess social media addiction. The BSMAS comprises six items. Each item is rated on a scale from one (very rarely) to five (very often). The items will be used to calculate the scores, with higher numbers indicating a higher degree of social media addiction. Demirci (2019) conducted the Turkish adaptation of the BSMAS used in this study. Demirci deemed the uni-dimensional structure of the Turkish BSMAS to be acceptable.
Fibromyalgia Impact Questionnaire (FIQ) | Baseline
  The Fibromyalgia Impact Questionnaire (FIQ) is a tool designed to assess and evaluate the status, progress and outcomes of individuals living with fibromyalgia (FM).
  It takes approximately five minutes to complete the FIQ, which is a self-administered instrument. The instructions are straightforward and the scoring is self-explanatory.
  The FIQ comprises 10 items. A 4-point Likert scale is used to rate the 11 questions in the first item, which are all related to physical functioning.
  Scores range from 0, indicating no impairment, to 10, indicating maximum impairment.

SECONDARY OUTCOMES:
Fear of Missing Out Scale (FOMOS) | Baseline
  The Fear of Missing Out Scale (FOMOS) will be used to assess fear of missing out. The FOMOS includes ten items. Each item is rated on a scale from one (not at all true) to five (absolutely true). The items will be summed, and higher scores will indicate a greater level of fear of missing out.
  The Turkish adaptation of the FOMOS used in this study was carried out by Can and Satici. The Turkish FOMOS's unidimensional structure was found to have acceptable fit indices, according to Can and Satici.
The Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a well-known tool used to assess sleep quality. It has been shown to be a reliable and valid measure, with adequate psychometric properties when used with adults. The PSQI is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in people who are being treated for health problems.
  Scores for each component range from 0 (no difficulty) to 3 (severe difficulty), and the sum of these scores produces a global score ranging from 0 to 21, with higher values indicating poorer sleep quality. A PSQI score greater than 5 is considered an indication of poor sleep quality, given its high sensitivity and specificity in identifying patients with sleep complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Ender Salbas, asst. proff., Principal Investigator — Balikesir University
Locations (1):
- Usak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Research data supporting this publication are available upon request from the authors. The datasets generated and/or analyzed during the current study are available from the corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the study was published
Access Criteria: If the study is published in a journal, then the data will be open

REFERENCES:
- [Result] Can G, Satici SA. Adaptation of fear of missing out scale (FoMOs): Turkish version validity and reliability study. Psicol Reflex Crit. 2019 Jan 22;32(1):3. doi: 10.1186/s41155-019-0117-4. PMID 32026206